CLINICAL TRIAL: NCT05501327
Title: A Randomized, Within Subject Controlled, Dose Regimen Study of SLI-F06 in Healthy Volunteers for Improvement in Scar Appearance
Brief Title: Dose Regimen Study of SLI-F06 in Healthy Volunteers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Scarless Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLI-F06-002
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Scar; Wound Healing
Keywords: Scar; Scar Appearance; Wound Healing
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Injection of SLI-F06 on Treatment Day 0, immediately after wound closure:
  * Formulation buffer (control)
  * 3.75 mg SLI-F06 total dose per wound (1X)
  * 7.5 mg SLI-F06 total dose per wound (2X)
  * 15 mg SLI-F06 total dose per wound (4X)
  Interventions: Drug: SLI-F06
- Cohort B (Experimental): Injection of SLI-F06 on Treatment Day 0, immediately after wound closure and on Days 1, 2, 3, 4:
  * Formulation buffer (control)
  * 3.75 mg SLI-F06 total dose per wound (1X)
  * 7.5 mg SLI-F06 total dose per wound (2X)
  * 15 mg SLI-F06 total dose per wound (4X)
  Interventions: Drug: SLI-F06
- Cohort C (Experimental): Injection of SLI-F06 on Treatment Day 0, immediately after wound closure and then 3 hours after for wounds dosed twice:
  * Formulation buffer (control) once
  * 7.5 mg SLI-F06 total dose per wound (2X) once
  * 3.75 mg SLI-F06 dose per wound (1X) twice, total dose 7.5 mg
  * 7.5 mg SLI-F06 total dose per wound (2X), total dose 15 mg
  Interventions: Drug: SLI-F06

INTERVENTIONS:
Drug: SLI-F06 — Skin injection of SLI-F06 at each wound edge after closure of punch biopsy excision.

SUMMARY:
Multi-center, dose-regimen, double-blind study evaluating the safety and efficacy of 4 doses of SLI-F06 compared with vehicle for improvement in scar appearance

DETAILED DESCRIPTION:
The is a Phase IIa dose-regimen study of small punch biopsy scars created on the upper and lower back of healthy patients. All excisions will be randomized to treatment with vehicle or 4 doses of SLI-F06 drug product. Patients will be divided into 3 cohorts, with Cohort B receiving the same doses as Cohort A but daily for a total of 5 days. Cohort C will receive up to twice the concentration of Cohort A potentially divided into 2 doses, with both cohorts treated only on treatment Day 0. Scars will be assessed for improvement by both the investigator and the patient at follow-up visits over 6-9 months.

Duration of study-approximately 7-10 months.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects, male or female, ages 18 to 65
2. Subjects with a Body Mass Index (BMI) 18.5-30 and at least 40 kg
3. Subjects with symmetrically located right and left scapular lines relative to the midline, and at least 12 cm distance between the right and left scapular lines.
4. Be able to follow study instructions and likely to complete all required visits.
5. Sign the Institutional Review Board (IRB)-approved informed consent form (ICF, which includes the Photographic and Video Release Form) prior to any study-related procedures being performed.

Exclusion Criteria:

1. Female subjects who are pregnant, breast-feeding, or of childbearing potential and not practicing reliable birth control methods
2. Subjects who were previously treated with SLI-F06
3. Subjects with evidence of hypertrophic or keloid scarring
4. Subjects with obvious back abnormalities (e.g., severe scoliosis)
5. Subjects with tattoos or previous scars in the study areas
6. Subjects who are poor surgical candidates

   1. Active disease that could interfere with or limit wound healing (e.g., diabetes, anemia, renal disease, hepatic disease, cardiac disease, or immune system disorders)
   2. History of clinically significant bleeding disorder or coagulation disorders
   3. Use of any tobacco/inhaled nicotine products including vaping within 12 months.
7. Subjects with evidence of skin infection or rash on the back
8. Subjects with history of active or uncontrolled skin disease (e.g., psoriasis, eczema, rosacea, vitiligo, skin cancer) that could interfere with the study or interpretation of the study outcomes
9. Subjects with a history of clinically significant allergies, especially drug hypersensitivity to lignocaine or allergy to adhesive surgical dressings
10. Subjects with any clinically significant abnormality following review of pre-study laboratory data and full physical examination
11. Subjects who are taking or have taken known anticoagulants:

    1. Blood thinners (e.g., coumadin, rivaroxaban, apixaban) within 2 months prior to day 0
    2. Others such as aspirin or aspirin containing products, Non-steroidal anti-inflammatory drugs (NSAIDs), vitamin E, fish oil within 14 days prior to day 0.
12. Subjects taking systemic or topical steroids within 4 weeks of Day 0
13. Subjects with excessive alcohol use, defined as >28 units of alcohol per week (1unit = 8 g alcohol, 1shot spirits, half- pint beer, or 5 oz wine)
14. Subjects who have evidence of drug abuse
15. Subjects who are known to have or had serum hepatitis or who are carriers of the hepatitis B surface antigen per medical history
16. Subjects with a history of poor or delayed wound healing (e.g., prior wound dehiscence, chronic wound, leg ulcer)
17. Subjects treated with an investigational drug or device within 30 days prior to day 0
18. Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, or may significantly interfere with the subject's participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2024-07-25 (Estimated); Study Completion 2024-10-25 (Estimated)

PRIMARY OUTCOMES:
Change in Scarless Labs Observer Scale | Months 1,3,6 and possibly 9
  Exploratory scale for observer to assess different scar parameters, including Surface Area, Elevation / Depression, Relief, Thickness, Pliability, Vascularity and Pigmentation. The observer then makes an Overall global assessment (scale 0 to -3) of the scar based on the clinical assessment of the scar parameters. All parameters are assessed on a scale of 0-3 (except pigmentation, -3 [hypo] to +3 [hyper]), where 0 correlates to a scar that is indistinguishable from normal skin with greater deviation from 0 correlating with more severe scar. The observer creates a forced rank between scars on the upper and lower back based on best (1) to worst (4) cosmetically.

SECONDARY OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) Observer Scale | Months 1,3,6 and possibly 9
  Established scar scale with observer rating of 1 (normal skin) to 10 (worst scar imaginable) for 6 different parameters (vascularity, pigmentation, thickness, relief, pliability, surface area) and overall opinion rated on the same 1-10 scale. The sum of these scores is added for a total value with a higher number being worse.
Scarless Labs Patient Scale | Months 1,3,6 and possibly 9
  Exploratory scale for subjects to assess different scar parameters, with 0 being no difference in pain or itching of the scar compared with normal skin and -3 being severe or worse. Patients then select a face on a modified Wong-Baker scale for their overall opinion of the scar.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth J Leeflang, MD, Study Director — Scarless Laboratories, Inc.
Locations (2):
- United States (2):
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - DermResearch, Austin, Texas

IPD SHARING:
Plan to Share IPD: No